CLINICAL TRIAL: NCT03010787
Title: A Four Part, Phase 1, First Time in Human, Single Centre Study in Healthy Male Subjects, Patient Volunteers With Crohn's Disease and in Healthy Patient Volunteers With a Terminal Ileostomy
Brief Title: A First Time in Human Study in Healthy Volunteers and Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VHsquared Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: V56501
Record Dates: First submitted 2016-12-12; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1 (Experimental): Single ascending dose of oral V565
  Interventions: Drug: V565
- Part 2 - V565 (Experimental): Single dose level of oral V565 TID for 14 days
  Interventions: Drug: V565
- Part 1 and 2 - placebo (Placebo Comparator): Oral placebo single dose (Part 1) or TID for 14 days (Part 2)
  Interventions: Drug: Placebo
- Part 3 (Experimental): Single dose of V565 in patient volunteers
  Interventions: Drug: V565
- Part 4 (Experimental): Single ascending dose of V565 in patients with Crohn's Disease
  Interventions: Drug: V565

INTERVENTIONS:
Drug: V565 — single ascending dose of V565
  Arms: Part 1
Drug: V565 — Multiple dose
  Arms: Part 2 - V565
Drug: Placebo — Single and multiple dose
  Arms: Part 1 and 2 - placebo
Drug: V565 — Open-label single dose
  Arms: Part 3
Drug: V565 — Open-label single ascending dose
  Arms: Part 4

SUMMARY:
A multi-part study to investigate the safety, tolerability and local and systemic pharmacokinetics of V565

ELIGIBILITY:
Inclusion Criteria:

* Parts 1 and 2

  1. Adult male subjects aged 18 to 45 years inclusive.
  2. Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive.
  3. Body weight between 50.0 and 100.0 kg inclusive.
  4. Subjects who are healthy as determined by pre study medical history, physical examination and 12-lead ECG, and clinical laboratory tests
* Part 3

  1. Adult male or female subjects aged 18 to 65 years.
  2. Ileostomy for a minimum of 18 months for a non malignant disease indication.
  3. A BMI between 18.0 and 32.0 kg/m2 inclusive.
  4. Body weight between 50.0 and 100.0 kg inclusive.
  5. Subjects who are healthy as determined by pre study medical history, physical examination and 12-lead ECG, and clinical laboratory tests
* Part 4

  1. Adult male or female subjects aged 18 to 65 years.
  2. A confirmed diagnosis of Crohn's disease for a minimum of 6 months.
  3. A BMI between 15.0 and 32.0 kg/m2 inclusive.
  4. Subjects who have no other significant co-morbidity (other than those associated with Crohn's disease).
  5. Subjects whose medical history, physical examination, clinical laboratory test results and 12-lead ECG have no clinically relevant abnormalities (other than those associated with Crohn's disease).

Exclusion Criteria:

* Parts 1 and 2

  1. A clinically significant abnormal medical history or clinically significant abnormal physical examination, including history of febrile illness within 1 week prior to the first dose.
  2. A history of severe allergies, non-allergic drug reactions, or multiple drug allergies.
  3. A known hypersensitivity to TNF inhibitors or any of the inactive ingredients of the study treatment.
  4. A history of significant gastrointestinal (GI) disease, including GI motility disorders, GI malignancy or of polyposis coli.
  5. Previous surgery to the GI tract with the exception of appendectomy.
  6. A history of malignancy.
  7. Any other condition which in the investigator's opinion will interfere with the trial or interpretation of the results.
* Part 3

  1. A history of Crohn's disease.
  2. A clinically significant abnormal medical history (other than the condition leading to ileostomy) or clinically significant abnormal physical examination, including history of febrile illness within 1 week prior to the first dose.
  3. A history of severe allergies, non-allergic drug reactions, or multiple drug allergies.
  4. A known hypersensitivity or contraindication to TNF inhibitors or any of the inactive ingredients of the study treatment.
  5. A known history of heart disease.
  6. Any clinical evidence of active inflammatory bowel disease.
  7. Any other condition which in the investigator's opinion will interfere with the trial or interpretation of the results.
* Part 4

  1. Subjects with severe Crohn's disease such as: those requiring surgery; those with a current abscess; those with a non inflammatory stricture; those with a history of obstruction.
  2. Having ever received anti-TNF-α therapy or other biologics.
  3. Required an increase in dose of either steroids or immunosuppressant therapy within the past 6 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability: treatment-emergent AEs including clinically significant changes in physical examinations, safety lab tests, ECGs or vital signs | Up to 14 days
Measurement of the concentrations of V565 in ileal fluid following a single dose | 24 hours

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of V565: Cmax | 72 hours
Evaluation of pharmacokinetic parameter of V565: AUC | 72 hours
Evaluation of pharmacokinetic parameter of V565: tmax | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Nurbhai, MBChB, Study Director — VHsquared Ltd.
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, Quintiles Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No